CLINICAL TRIAL: NCT06124755
Title: Comparing the Efficacy of Heparin-boned Viabahn@ Endoprosthesis and Paclitaxel-coated Balloons for Endovascular Treatment of Complex Femoropopliteal Lesions
Brief Title: The Efficacy of Heparin-boned Viabahn Endoprosthesis and Paclitaxel-coated Balloons for Complex Femoropopliteal Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Chengdu University of Traditional Chinese Medicine (Other); Second Affiliated Hospital of Soochow University (Other); First Affiliated Hospital of Zhejiang University (Other); Xuanwu Hospital, Beijing (Other); Qingdao Haici Hospital (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Fudan University (Other); Huashan Hospital (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The Virtue study
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Viabahn endoprosthesis; Drug-coated balloon
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viabahn endoprosthesis group (Experimental): Femoropopliteal lesions treated with Viabahn endoprosthesis.
  Interventions: Device: Viabahn endoprosthesis group
- Drug-coated balloon group (Active Comparator): Femoropopliteal lesions treated with drug-coated balloon endoprosthesis.
  Interventions: Device: Drug-coated balloon group

INTERVENTIONS:
Device: Viabahn endoprosthesis group — Patients underwent endovascular treatment for femoropopliteal lesions. The lesion will be treated by Viabahn endoprosthesis.
  Arms: Viabahn endoprosthesis group
Device: Drug-coated balloon group — Patients underwent endovascular treatment for femoropopliteal lesions. The lesion will be treated by drug-coated balloon.
  Arms: Drug-coated balloon group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the Viabahn endoprosthesis for treating long femoropopliteal lesions (stenosis ≥ 25cm, occlusion ≥ 15cm) or recurrent in-stent restenosis compared to drug-coated balloons (DCB) with or without a bailout bare nitinol stent.

DETAILED DESCRIPTION:
This is a multicenter, prospective, 1:1 randomized clinical trial with clinical and image follow-up for two years post-procedure. Approximately 60 subjects will be enrolled and randomized into a Viabahn preferred group (study arm) or drug-coated balloons (DCB) group (control arm); Each group will include 30 patients. All enrolled patients will be followed up for 12 months to assess the incidence of restenosis by duplex ultrasound and major adverse events. Follow-up visits occur at 12 and 24 months, as well as telephone visits after 1, 6, 9 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. The patient presented a score from 2 to 5 following Rutherford classification.
2. The patient is willing to comply with specified follow-up evaluations at the specified times.
3. The patient is ≥ 18 years old.
4. Patient understands the nature of the procedure and provides written informed consent before enrolment in the study
5. The patient has a projected life expectancy of at least 24 months
6. Before enrolment, the guidewire has crossed the target lesion
7. Subject has a de novo or restenotic lesion with ≥ 70% stenosis in femoropopliteal artery, and for de novo lesion, the total lesion length ≥ 25cm, or chronic total occlusion (CTO) length ≥15cm.
8. There is angiographic evidence of patent infrageniculate popliteal artery and at least one distal runoff to the foot.
9. Origin and proximal 1 cm of Superficial Femoral Artery (SFA) are patent.
10. Reference vessel diameter (RVD) ≥ 4 mm by visual estimation.

Exclusion Criteria:

1. Previous bypass surgery or stenting in the target vessel
2. Patients who exhibit acute intraluminal thrombus at the target lesion vessel
3. Patients with known hypersensitivity or contraindication to any of the following medications: Nitinol-titanium, antiplatelet therapy, anticoagulants, or thrombolytics therapy
4. Pregnant women or Female patients with potential childbearing
5. Use of thrombectomy, atherectomy, or laser devices during the procedure
6. Untreated inflow disease of the ipsilateral pelvic arteries (more than 50% stenosis or occlusion)
7. The patient is currently participating in another investigational drug or device study that interferes with the study
8. Significant renal dysfunction (Serum creatinine >3.0mg/dl)
9. Patient with Known allergy to contrast media
10. Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of anti-platelet therapy.
11. Femoral or popliteal aneurysm.
12. Current peritoneal or hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 24-month
  Peak systolic velocity ratio (PSVR ≤2.4) without any repeat intervention.
Freedom from a composite of Major adverse events (MAEs) | 24-month
  Freedom from MAEs is defined as freedom from clinically-driven target vessel revascularization (CD-TVR), major amputation, and all-cause of death

SECONDARY OUTCOMES:
Procedural success | Immediately after interventional surgery
  Procedural success is defined as technical or device success without major adverse events during the hospital stay.
Primary assisted patency | 24-month
  Primary assisted patency is defined as maintaining patency in the target vessel after a repeat intervention to regain patency prior to complete occlusion.
Secondary patency | 24-month
  Secondary patency is defined as maintaining patency in the target vessel after a repeat intervention to correct complete occlusion in the treated arterial segment.
Clinically-driven target vessel revascularization (CD-TVR) | 24-month
  clinically-driven target vessel revascularization (CD-TVR) is defined as repeat intervention performed during enrollment in the clinical study.
Primary sustained clinical improvement | 24-month
  Defined as a sustained upward shift of at least one category on the Rutherford classification without the need for repeated target lesion revascularization (TLR) in surviving patients.
Secondary sustained clinical improvement | 24-month
  Defined as a sustained upward shift of at least one category on the Rutherford classification3, including the need for repeated target lesion revascularization (TLR) in surviving patients.
Vasc quality of life score | 24-month
  Change of Vasc quality of life score

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China